CLINICAL TRIAL: NCT06628037
Title: A Phase 1 Maximum Tolerated Dose Study of SN514-066b in Adult Patients With Deep Partial Thickness Dermal Burns
Brief Title: SN514-066b Enzyme in Deep Partial Thickness Burns
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SERDA bv (Industry)
Collaborators: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRDA-SN514-102
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Burn Injury
Keywords: Maximum tolerated dose; Debridement
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1st cohort (Experimental): Testing 0.10% SN514-066b gel
  Interventions: Biological: SN514-066b
- 2nd cohort (Experimental): Testing 0.20% gel
  Interventions: Biological: SN514-066b
- 3rd cohort (Experimental): Testing 0.40% gel
  Interventions: Biological: SN514-066b
- 4th cohort (Experimental): Testing 0.80% gel
  Interventions: Biological: SN514-066b

INTERVENTIONS:
Biological: SN514-066b — Enzyme debrider

SUMMARY:
This study will examine the tolerability of a gel formulation of the enzyme SN514 in patients with burns suitable for enzymatic debridement. In a rising dose fashion by sequential cohort, concentrations of 0.1%, 0.2%, 0.4% and 0.8% will be tested. Groups of 3 will undergo daily debridement for up to 7 days. Extent of debridement and adverse signs and symptoms will be recorded daily. Dose escalation will stop if a dose level is found to be intolerable. Dose escalation may accelerate if a tested dose is entirely ineffective. There is no placebo control as all burn wounds require debridement.

DETAILED DESCRIPTION:
The design of the study is a sequential rising dose to the maximum tolerated dose, in which each subject will be exposed to only one concentration of the test article. Dose limiting toxicities are defined as "Severe" or CTCAE v5 Grade 3 or higher adverse events. This study in burn patients is designed to apply SN514-066b over 25 cm2 (0.14% TBSA for a 1.73 m2 adult) up to 500 cm2 (2.9%), at sequentially rising concentrations of 0.1%, 0.2%, 0.4% and 0.8% (< 1.0 mg/cm2). The highest exposure would be 0.8% (8 g per 100 cc of gel) over 2.9% of 1.73 m2 = 800 mg or 11.4 mg/kg applied topically (70 kg patient).

ELIGIBILITY:
Main Inclusion Criteria:

1. Thermal burns caused by fire/flame, scalds or contact
2. Total burns area available for treatment is 25 to 500 cm2 (a larger area may be burned, but the treatment area must be limited to the stated size, and the treatment area must be exclusive of face, hands, genitalia and sites deemed to be at high risk for developing compartment syndrome)
3. Target burns for treatment is deep partial thickness (DPT) in depth

Main Exclusion Criteria:

1. Subject has another life threatening traumatic injury
2. Patient's proposed study wound site has any of the following conditions:

   * Electrical or chemical etiology
   * Pre-enrollment escharotomy
   * Area is devoid of circulation
   * Located on the face, perineum or genitalia
   * Clinical evidence of wound infection
3. Poorly controlled diabetes mellitus (HbA1c >12%)
4. BMI greater than 40 kg/m2
5. Cardio-pulmonary disease (MI within 6 months prior to injury, severe or unstable ischemic heart disease, severe or unstable heart failure, severe pulmonary hypertension, severe COPD or pre-existing oxygen-dependent pulmonary diseases, severe broncho-pneumonia within 1 month prior to injury, steroid dependent asthma, or uncontrolled asthma)
6. Pre-existing diseases which interfere with circulation (severe peripheral vascular disease, severe circulatory edema and/or lymphedema, regional lymph nodes dissection, significant varicose veins)
7. Any conditions that would preclude safe treatment or adding further risk to the basic acute burn trauma (such as severe immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder, severe cardiovascular disorder, significant pulmonary disorder, significant liver disorder including post alcoholic abuse impaired function or neoplastic disease, blast injury)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated concentration of SN514 gel when applied topically to deep partial thickness burn wounds | Daily x 7days
  Number of participants with treatment-related adverse events of Grade 3 or higher as assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, where a higher grade on the scale of 1 to 5 is a worse outcome.

SECONDARY OUTCOMES:
Evaluate the time course and extent of debridement when applied daily for up to 7 days | Daily x 7days
  Percent of eschar removed following each 24 hr debridement
Evaluate effects of treatment on inflammation | Daily x 7days
  Changes from baseline to end of treatment in blood levels of C-reactive protein (CRP) in mg/dL, serum tryptase in ng/mL, and total complement activity (CH50) level in hemolytic units.
Observe the incidence of wound erythema | Daily x 7days
  Record daily the appearance of new, spreading or darkening redness of the treated or adjacent tissue
Incidence of wound purulence | Daily for 7 days
  Observe daily for the appearance of purulent material in the treatment area

CONTACTS AND LOCATIONS:
Locations (1):
- USAISR Burn Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a single center trial. If a subsequent burn study is conducted, then certain data may be shared with future investigators. All data are submitted to the IND.